CLINICAL TRIAL: NCT02477605
Title: Clinical Comparison of 27+® and 23-gauge ULTRAVIT® 7500 Cpm Vitrectomy Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VRH172-P001
Record Dates: First submitted 2015-06-18; First posted 2015-06-23 (Estimated); Results first posted 2017-07-27 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-06

CONDITIONS: Vitreoretinal Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 27-gauge pak (Experimental): CONSTELLATION® 27-gauge combined surgical pak used during vitrectomy surgery
  Interventions: Device: CONSTELLATION® 27-gauge Combined Surgical Pak; Procedure: Vitrectomy surgery
- 23-gauge pak (Active Comparator): CONSTELLATION® 23-gauge combined surgical pak used during vitrectomy surgery
  Interventions: Device: CONSTELLATION® 23-gauge Combined Surgical Pak; Procedure: Vitrectomy surgery

INTERVENTIONS:
Device: CONSTELLATION® 27-gauge Combined Surgical Pak — Sterile single-use supplies necessary to perform 1 vitrectomy surgery: 1 ULTRAVIT® 27-gauge 7500 cuts per minute (cpm) vitrectomy probe and a 27-gauge EDGEPLUS® Valved Entry System comprised of 3 trocar/cannulas and related accessories.
  Arms: 27-gauge pak
Device: CONSTELLATION® 23-gauge Combined Surgical Pak — Sterile single-use supplies necessary to perform 1 vitrectomy surgery: 1 ULTRAVIT® 23-gauge 7500 cuts per minute (cpm) vitrectomy probe and a 23-gauge EDGEPLUS® trocar/cannula set comprising of 3 trocars/cannulas and related accessories.
  Arms: 23-gauge pak
Procedure: Vitrectomy surgery — Microincisional pars plana vitrectomy (PPV) surgery for the treatment of various vitreoretinal diseases ranging from simple to advanced cases

SUMMARY:
The purpose of this study is to compare the treatment day change between immediate postoperative and immediate preoperative intraocular pressure (IOP) between 27-gauge and 23-gauge vitrectomy instruments.

DETAILED DESCRIPTION:
Required follow-up for this study is 3 months post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent and attend all required study visits;
* Requires vitrectomy in at least one eye;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Previous vitrectomy or glaucoma surgery;
* Planned treatment requires scleral buckling, combined procedures (eg, cataract surgery), silicone oil, and expansive gas other than sterile air;
* Treated with topical IOP lowering medication(s) at any time from baseline assessment to time of surgery;
* Pregnant or planning to become pregnant during the course of the trial;
* Other protocol-defined exclusion criteria may apply.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2015-07-16 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Manager, Surgical, GCRA, Study Director — Alcon, A Novartis Division
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 6 study centers located in the US.
Pre-assignment Details: Of the 137 enrolled, 1 subject was exited as a screen failure prior to randomization. This reporting group includes all randomized subjects (136).
Groups:
- 27-Gauge: CONSTELLATION® 27-gauge combined surgical pak used during vitrectomy surgery
- 23-Gauge: CONSTELLATION® 23-gauge combined surgical pak used during vitrectomy surgery
Period: Overall Study
Arm/Group | 27-Gauge | 23-Gauge
Started | 68 | 68
Randomized and Treated | 67 | 68
Completed | 67 | 64
Not Completed | 1 | 4
Not completed — Discontinued prior to treatment | 1 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Administered gas during surgery | 0 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized subjects (Intent-to-Treat Analysis Set).
Groups:
- Total: Total of all reporting groups
Arm/Group | 27-Gauge | 23-Gauge | Total
Number analyzed (Participants) | 68 | 68 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (11.55) | 67.0 (11.65) | 66.4 (11.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 45 | 88
  Male | 25 | 23 | 48

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Intraocular Pressure (IOP) on Operative Day
Description: IOP (fluid pressure inside the eye) was assessed using the study specified tono-pen and measured in millimeters of mercury (mmHg). Change was defined as the difference between immediate postoperative IOP and immediate preoperative IOP. A greater change in IOP may indicate a less stable posterior chamber and/or a more invasive surgery.
Time Frame: Day 0 preoperative, Day 0 postoperative
Population: Intent-to-Treat Analysis Set. Number Analyzed is the number of subjects with data.
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | 27-Gauge | 23-Gauge
Number analyzed (Participants) | 67 | 68
mmHG | -0.40 (6.603) | -3.05 (7.639)

2. Secondary Outcome: Mean Conjunctival Edema Score at Week 1
Description: Conjunctival edema (swelling) was assessed during examination by the investigator and graded on a scale of 0-3, where 0=Absent and 3=Severe. Each sclerotomy wound was graded as infusion, vitrectomy probe, and illuminator and the average of the three was the overall Conjunctival Edema Score at the visit. Only one eye (study eye) contributed to the analysis.
Time Frame: Week 1 post operative
Population: Intent-to-Treat Set. Number Analyzed is the number of subjects with data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 27-Gauge | 23-Gauge
Number analyzed (Participants) | 67 | 67
units on a scale | 0.02 (0.124) | 0.10 (0.246)

3. Secondary Outcome: Mean Post-operative Pain Rating at Day 1
Description: The subject was asked to rate post-operative pain in the study eye using a score of 0-10, where 0=no pain and 10=the worst pain imaginable.
Time Frame: Day 1 post operative
Population: Intent-to-Treat Analysis Set. Number Analyzed is the number of subjects with data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 27-Gauge | 23-Gauge
Number analyzed (Participants) | 67 | 67
units on a scale | 0.9 (1.75) | 0.6 (1.20)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent for the duration of a subject's participation in the study (up to 4 months).
Description: An AE was defined as any untoward medical occurrence in a subject administered a clinical trial treatment (ie, implant with an investigational device) regardless of whether the event has a causal relationship with the treatment. AEs were obtained through solicited and spontaneous comments from subjects and observations by the Investigator. Safety analysis set included all subjects/eyes exposed to the investigational device. One subject randomized to 27-gauge was treated with 23-gauge instead.
Groups:
- 27-Gauge Treated Eye; 23-Gauge Treated Eye: Ocular events, treated (study) eye
- 27-Gauge Fellow Eye; 23-Gauge Fellow Eye: Ocular events, untreated (fellow) eye
- 27-Gauge Systemic; 23-Gauge Systemic: Non-ocular adverse events
Arm/Group | 27-Gauge Treated Eye | 27-Gauge Fellow Eye | 27-Gauge Systemic | 23-Gauge Treated Eye | 23-Gauge Fellow Eye | 23-Gauge Systemic
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/66 | 0/66 | 0/69 | 0/69 | 0/69
Serious Adverse Events (participants affected / at risk) | 15/66 | 0/66 | 0/66 | 16/69 | 0/69 | 1/69
Other Adverse Events (participants affected / at risk) | 18/66 | 0/66 | 0/66 | 14/69 | 0/69 | 0/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 27-Gauge Treated Eye (N=66) | 27-Gauge Fellow Eye (N=66) | 27-Gauge Systemic (N=66) | 23-Gauge Treated Eye (N=69) | 23-Gauge Fellow Eye (N=69) | 23-Gauge Systemic (N=69)
Cataract (Eye disorders) | 7 (7) | 0 (0) | 0 (0) | 9 (9) | 0 (0) | 0 (0)
Hypotony of eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Macular fibrosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 2 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Retinopathy proliferative (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 6 (6) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraocular pressure decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Craniotomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye laser surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Retinal laser coagulation (Surgical and medical procedures) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Vitrectomy (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 27-Gauge Treated Eye (N=66) | 27-Gauge Fellow Eye (N=66) | 27-Gauge Systemic (N=66) | 23-Gauge Treated Eye (N=69) | 23-Gauge Fellow Eye (N=69) | 23-Gauge Systemic (N=69)
Conjunctival haemorrhage (Eye disorders) | 9 (9) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0)
Conjunctival oedema (Eye disorders) | 6 (6) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 0 (0)
Punctate keratitis (Eye disorders) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 6 (7) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.